CLINICAL TRIAL: NCT05368090
Title: Endoscopic Ultrasound-guided Radiofrequency Ablation as a Novel Treatment Option Compared With Adrenalectomy in Left-sided Primary Aldosteronism
Brief Title: Endoscopic Ultrasound-guided Radiofrequency Ablation in Primary Aldosteronism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 422376
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Primary Aldosteronism; Aldosterone-Producing Adenoma; Hypercortisolism
Keywords: radio frequency ablation; postoperative hypoaldosteronism; postoperative hypocortisolism; metabolic comorbidity
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma; Cushing Syndrome

STUDY DESIGN:
Intervention Model Description: Four EUS-RFA intervention study groups Group 1: PA with lateralisation to left adrenal and left-sided tumour for EUS-RFA Group 2: PA with suspected left-sided overweight of aldosterone overproduction but not AVS-verified left-sided lateralisation for EUS-RFA as "debulking" procedure Group 3: MACS with unilateral tumour in the left adrenal and unilateral cortisol overproduction verified by AVS, for EUS-RFA Group 4: MACS with bilateral adrenal tumours and AVS-verified bilateral cortisol overproduction for EUS-RFA as "debulking" procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EUS-RFA of PA with AVS-verified left lateralisation (Experimental): PA patients with AVS-confirmed lateralisation to the left adrenal and signed study consent will be included in this study group. EUS will be performed. If EUS identifies an adrenal nodule in the left adrenal, EUS-guided fine needle tissue sampling of the adenoma will be performed, before a subsequent EUS-RFA treatment procedure will be performed. Follow-up after 2 weeks, 3 months and 12 months for evaluation of clinical and biochemical outcome, and procedural complications.
  Interventions: Procedure: EUS-RFA of left adrenal tumour in PA with AVS-verified left lateralisation
- EUS-RFA of PA without verified left lateralisation, for aldosterone "debulking" (Experimental): PA patients with suspicion of aldosterone overproduction in their left adrenal, but without fulfilling the strict AVS lateralization criteria, either due to a non-representative AVS, or a representative AVS but without significant left-sided lateralization (LI < 4), and where the study investigators consider EUS-RFA treatment as an aldosterone-reducing procedure to be of high potential clinical and biochemical benefit for the patient, will be included in this study group after signed consent. EUS will be performed. If EUS identifies an adrenal nodule in the left adrenal, an EUS-guided fine needle tissue sampling of the adenoma will be performed, before a subsequent EUS-RFA treatment procedure. Follow-up after 2 weeks, 3 months and 12 months for evaluation of clinical and biochemical outcome, and procedural complications.
  Interventions: Procedure: EUS-RFA of left adrenal tumour in PA, "debulking group"
- EUS-RFA of MACS with left lateralisation and left adrenal tumour (Experimental): MACS patients with AVS-confirmed lateralisation the left adrenal gland and CT showing left-sided tumour will be included in this study group after signed consent. EUS will be performed, and a EUS-guided fine needle tissue sampling of the adenoma will be performed, before a subsequent EUS-RFA treatment procedure. Follow-up after 2 weeks, 3 months and 12 months for evaluation of clinical and biochemical outcome, and procedural complications.
  Interventions: Procedure: EUS-RFA of left adrenal tumour in MACS with AVS-verified left lateralisation
- EUS-RFA of MACS with bilateral cortisol overproduction and bilateral tumours (Experimental): MACS patients with AVS-confirmed bilateral cortisol overproduction and bilateral tumours will be included in this study group after signed study consent. EUS will be performed, and EUS-guided fine needle tissue sampling of the adenoma will be performed, before a subsequent EUS-RFA treatment procedure. Follow-up after 2 weeks, 3 months and 12 months for evaluation of clinical and biochemical outcome, and procedural complications.
  Interventions: Procedure: EUS-RFA of left adrenal tumour in MACS with bilateral overproduction, "debulking group

INTERVENTIONS:
Procedure: EUS-RFA of left adrenal tumour in PA with AVS-verified left lateralisation — Patients will fast, receive prophylactic antibiotics and conscious sedation prior to the endoscopic procedure.The procedure is performed with a standard linear echo-endoscope with a 3.7 mm or larger working channel. The left adrenal is identified from the fundus of the stomach. Color-Doppler is used to map adrenal vascularity. Ultrasound contrast is used to demarcate the border of the tumour. EUS-guided fine needle tissue sampling from tumour tissue is performed. The RFA ablation catheter is water-cooled and stable temperature is maintained at 70-75 degrees celsius until formation of heat bubbles can be seen on EUS. If necessary, the procedure is repeated after moving the probe until the whole adenoma volume is ablated. Ultrasound contrast medium is used after the procedure to ensure that the target for the ablation is non vascularized, before termination. The patients will be observed at the postoperative unit a few hours, and further in the ward for 24h
  Arms: EUS-RFA of PA with AVS-verified left lateralisation
Procedure: EUS-RFA of left adrenal tumour in PA, "debulking group" — Patients will fast, receive prophylactic antibiotics and conscious sedation prior to the endoscopic procedure.The procedure is performed with a standard linear echo-endoscope with a 3.7 mm or larger working channel. The left adrenal is identified from the fundus of the stomach. Color-Doppler is used to map adrenal vascularity. Ultrasound contrast is used to demarcate the border of the tumour. EUS-guided fine needle tissue sampling from tumour tissue is performed. The RFA ablation catheter is water-cooled and stable temperature is maintained at 70-75 degrees celsius until formation of heat bubbles can be seen on EUS. If necessary, the procedure is repeated after moving the probe until the whole adenoma volume is ablated. Ultrasound contrast medium is used after the procedure to ensure that the target for the ablation is non vascularized, before termination. The patients will be observed at the postoperative unit a few hours, and further in the ward for 24h
  Arms: EUS-RFA of PA without verified left lateralisation, for aldosterone "debulking"
Procedure: EUS-RFA of left adrenal tumour in MACS with AVS-verified left lateralisation — Patients will fast, receive prophylactic antibiotics and conscious sedation prior to the endoscopic procedure.The procedure is performed with a standard linear echo-endoscope with a 3.7 mm or larger working channel. The left adrenal is identified from the fundus of the stomach. Color-Doppler is used to map adrenal vascularity. Ultrasound contrast is used to demarcate the border of the tumour. EUS-guided fine needle tissue sampling from tumour tissue is performed. The RFA ablation catheter is water-cooled and stable temperature is maintained at 70-75 degrees celsius until formation of heat bubbles can be seen on EUS. If necessary, the procedure is repeated after moving the probe until the whole adenoma volume is ablated. Ultrasound contrast medium is used after the procedure to ensure that the target for the ablation is non vascularized, before termination. The patients will be observed at the postoperative unit a few hours, and further in the ward for 24h
  Arms: EUS-RFA of MACS with left lateralisation and left adrenal tumour
Procedure: EUS-RFA of left adrenal tumour in MACS with bilateral overproduction, "debulking group — Patients will fast, receive prophylactic antibiotics and conscious sedation prior to the endoscopic procedure.The procedure is performed with a standard linear echo-endoscope with a 3.7 mm or larger working channel. The left adrenal is identified from the fundus of the stomach. Color-Doppler is used to map adrenal vascularity. Ultrasound contrast is used to demarcate the border of the tumour. EUS-guided fine needle tissue sampling from tumour tissue is performed. The RFA ablation catheter is water-cooled and stable temperature is maintained at 70-75 degrees celsius until formation of heat bubbles can be seen on EUS. If necessary, the procedure is repeated after moving the probe until the whole adenoma volume is ablated. Ultrasound contrast medium is used after the procedure to ensure that the target for the ablation is non vascularized, before termination. The patients will be observed at the postoperative unit a few hours, and further in the ward for 24h
  Arms: EUS-RFA of MACS with bilateral cortisol overproduction and bilateral tumours

SUMMARY:
In this study, the investigators will perform endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) treatment of left-sided adrenal tumours in patients with primary aldosteronism (PA) and in patients with mild autonomous cortisol secretion (MACS). Four different study groups will all receive EUS-RFA of left-sided adrenal tumours. Clinical and biochemical outcome as well as procedural safety will be evaluated. In study patients with verified lateralised aldosterone or cortisol overproduction to the left adrenal, outcome will be compared with control groups performing conventional unilateral adrenalectomy.

Study group 1: PA patients with AVS-verified left sided lateralisation and a EUS-detectable tumour in the left adrenal for EUS-RFA treatment.

Study group 2: PA patient with suspected left-sided overweight of aldosterone production and a EUS-detectable tumour but without strict lateralisation of their aldosterone overproduction, for EUS-RFA treatment as an aldosterone "debulking" procedure.

Study group 3: patients with MACS with AVS-verified lateralisation of cortisol overproduction to the left adrenal and EUS-detectable tumour for EUS-RFA treatment Study group 4: patients with MACS with bilateral adrenal tumours and verified bilateral overproduction of cortisol for EUS-RFA treatment as a cortisol "debulking" procedure.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the most common cause of secondary hypertension, and is associated with worse cardiovascular outcome than primary hypertension. Early diagnosis and treatment is paramount to avoid excess morbidity and death. The two main forms of PA are unilateral PA, often caused by an aldosterone-producing adenoma (APA), and bilateral PA. Differentiation between unilateral and bilateral disease determines treatment options. Adrenal vein sampling (AVS) is the recommended procedure to determine PA subtype, unilateral or bilateral. For unilateral PA surgery with unilateral adrenalectomy is recommended treatment. For PA without fulfilling lateralisation criteria, life-long medical treatment is recommended.

Mild autonomous cortisol production (MACS) is present in 20-30% of all adrenal incidentalomas, and is associated with the metabolic syndrome (hypertension, diabetes, obesity and osteoporosis). Therefore these patients carry increased risk of developing cardiovascular disease. Optimal treatment is debated, and based on the degree of MACS, degree of metabolic complications, and the patient's own opinion. Unilateral adrenalectomy is an option if the overproduction is unilateral, but in 15 % of cases, the overproduction is bilateral, and treatment strategy even more troublesome.

The left adrenal is situated in near proximity to the stomach and is easily reached by endoscopic ultrasound (EUS), and may be targeted for RFA, treating an aldosterone- or cortisol-producing tumour only, and spearing the remaining adrenal. In this study we introduce EUS-RFA as a new treatment option in the following patient groups:

Study group 1: PA patients with AVS-verified left sided lateralisation and a EUS-detectable tumour in the left adrenal for EUS-RFA treatment.

Study group 2: PA patient with suspected left-sided overweight of aldosterone production and a EUS-detectable tumour but without strict lateralisation of their aldosterone overproduction, for EUS-RFA treatment as an aldosterone "debulking" procedure.

Study group 3: patients with MACS with AVS-verified lateralisation of cortisol overproduction to the left adrenal and EUS-detectable tumour for EUS-RFA treatment Study group 4: patients with MACS with bilateral adrenal tumours and verified bilateral overproduction of cortisol for EUS-RFA treatment, as a cortisol "debulking" procedure.

For all study groups, if CT scan shows an adrenal nodule to the left adrenal, nodule size must be < 40 mm and enhancement value must fulfill criteria for a benign adenoma. Patients consenting to the EUS-RFA will have a EUS performed. If EUS of the left adrenal identifies an adrenal nodule, a fine needle tissue sampling will be performed. Thereafter EUS-guided RFA procedure of the tumour will be performed. After RFA treatment, the fine needle tissue sampling will undergo morphological and functional characterisation, including application of specific imaging mass cytometry for detection of aldosterone- or cortisol producing cells.

Clinical and biochemical outcome after EUS-RFA will be evaluated by the international PASO-criteria (PA) or ENSAT/ECE criteria (MACS). In patients with lateralised PA or lateralised MACS, clinical and biochemical outcome and postoperative hypoaldosteronism or hypocortisolism will be compared with conventional unilateral adrenalectomy. Inn all patients, procedural safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria all groups

* Signed written informed consent
* If CT scan shows an adrenal nodule to the same adrenal as AVS lateralisation result: nodule size < 4 cm and enhancement criteria for adrenal adenoma (native hounsfield units < 10 or relative wash-out > 40% or absolute wash-out > 60%)

PA unilateral group inclusion criteria:

* Age 18 to 60 years
* PA diagnosis confirmed according to Endocrine Society PA Guideline criteria
* AVS lateralisation to left adrenal (lateralisation index ≥ 4,0)

PA "debulking" group inclusion criteria:

* Age 18 to 70 years
* PA diagnosis confirmed according to Endocrine Society PA Guideline criteria

MACS unilateral and debulking group inclusion criteria:

* Age 18 to 80 years
* MACS diagnosis confirmed according to ENSAT/ECE Guideline criteria
* AVS lateralisation to the left adrenal, and visible left adrenal tumor on CT scan OR bilateral overproduction of cortisol on AVS, and bilateral tumors/hyperplasia on CT scan (debulking)

Exclusion Criteria all groups:

* CT scan suspicion of adrenal malignancy
* Patient refusal to undergo either EUS-RFA or adrenalectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical outcome in PA after EUS-RFA | 1 year
  Biochemical outcome will be evaluated by international standardised "Primary aldosteronism surgery outcome" (PASO) criteria at follow-up visits after 3 and 1 year
Clinical outcome in PA after EUS-RFA | 1 year
  Clinical outcome will be evaluated by international standardised PASO criteria at follow-up visits after 1 year
Biochemical outcome in MACS after EUS-RFA | 1 year
  Biochemical outcome will be evaluated at follow-up visits after 3 and 1 year, evaluated by the international European Network for Study of Adrenal Tumour (ENSAT) /European Society of Endocrinology (ESE) criteria
Clinical outcome in MACS after EUS-RFA | 1 year
  Clinical outcome will be evaluated at follow-up visits after 3 and 1 year, evaluated by the international ENSAT/ESE criteria

SECONDARY OUTCOMES:
Number of participants with procedural complications of EUS-RFA compared with unilateral adrenalectomy | 3 months
  Procedural complications of EUS-RFA compared with unilateral adrenalectomy will be performed using the Clavien-Dindo classification.
Length of hospital stay after EUS-RFA compared with after adrenalectomy | 3 months
  Length of hospital stay after EUS-RFA will be compared with adrenalectomy, and will be evaluated at follow-up after 3 months
Number of participants with postoperative hypoaldosteronism | 3 months
  Number of participants with postoperative hypoaldosteronism after EUS-RFA will be compared with unilateral adrenalectomy by biochemical assessment at 3 months after treatment
Number of participants with postoperative hypocortisolism | 6 weeks
  Number of participants with postoperative hypocortisolism after EUS-RFA will be compared with unilateral adrenalectomy. In patients with an abnormal pre-treatment 1 mg dexamethasone suppression test or a low morning cortisol < 300 nmol/L after RFA or adrenalectomy, individual advise of cortisone acetate replacement therapy will be given and an stimulation adrenocorticotropic hormone (ACTH) test will be performed in the Endocrinology Out-patient clinic ~ 6 weeks of discharge
Change from baseline in health-related quality of life at 1 year | 1 year
  Change in health-related quality of life after treatment compared with pre-treatment, will be measured by the validated RAND-36 Health Survey, and will be compared in the EUS-RFA group and adrenalectomy group.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Grytaas, MD phd, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway